CLINICAL TRIAL: NCT02925377
Title: Efficacy of a Specific Warm-up Program to Improve Static and Dynamic Postural Control in Adult Female Handball Players
Brief Title: Neuromuscular Warm-up Intervention to Improve Postural Control in Female Handball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Prof. Dr., University of Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 115_15Bc
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Postural Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neuromuscular (Experimental): Neuromuscular warm-up
  Interventions: Behavioral: Neuromuscular warm-up
- Control (Active Comparator): Standard warm-up
  Interventions: Behavioral: Standard warm-up

INTERVENTIONS:
Behavioral: Neuromuscular warm-up — The intervention group replaced their regular warm-up routine with seven neuromuscular warm-up exercises performed for 15 minutes prior to each practice session (3x/week) over a period of eleven weeks.
  Arms: Neuromuscular
Behavioral: Standard warm-up — Athletes in the control group followed their regular 15 minutes warm-up routine provided by the team coaches.
  Arms: Control

SUMMARY:
Female handball athletes are at a particular risk of sustaining lower extremity injuries. The study examines time-dependent adaptations of static and dynamic balance as potential injury risk factors to a specific warm-up program focusing on neuromuscular control.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Female
* Handball players
* Actively participated in competitions
* Uninjured at study enrollment

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline: Static postural control | 3, 6, 9, and 11 weeks
  Postural sway (center of pressure sway velocity) during unipedal quiet standing, eyes opened (20 seconds)
Change from Baseline: Dynamic postural control | 3, 6, 9, and 11 weeks
  Star Excursion Balance Test (SEBT)

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Zech, Prof. Dr., Principal Investigator — Institute of Sports Science, Friedrich-Schiller-Universität Jena
Locations (1):
- Institute of Sport Science and Sport; FAU Erlangen-Nürnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Steib S, Zahn P, Zu Eulenburg C, Pfeifer K, Zech A. Time-dependent postural control adaptations following a neuromuscular warm-up in female handball players: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2016 Oct 13;8:33. doi: 10.1186/s13102-016-0058-5. eCollection 2016. PMID 27757240